CLINICAL TRIAL: NCT06174870
Title: The Effect of Inspiratory Muscle Training on Blood Pressure and Functional Capacity in Elderly With Hypertension
Acronym: IMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Phayao (Other)
Responsible Party: Principal Investigator, EAKARACH WONGSAYA, Lecturer, University of Phayao
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPhayao
Record Dates: First submitted 2023-12-01; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Elderly; Hypertension
Keywords: Elderly; Hypertension; Inspiratory muscle training
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group
- Intervention (Experimental): IMT group
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — Inhale against 60% of Maximal inspiratory pressure 30breaths/day 5days/week for 6 weeks
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to investigate in elderly with hypertension . The main question it aim to answer is:

• Investigate the effect of inspiratory muscle training on inspiratory muscle strength, blood pressure and physical capacity

Participants will be random in to 2 group and measure baseline. Control group will advise to maintain normal daily life activity. and Intervention group will receive inspiratory muscle training (IMT) with 60% of Maximal inspiratory pressure. Intervention group will perform IMT 30 breaths/day, 5 days a week for 6 weeks.

after 6 weeks both group will remeasure variable again as post test

ELIGIBILITY:
Inclusion Criteria:

* Elderly with hypertension
* BMI 18.5 - 29.9 kg/m2

Exclusion Criteria:

* Unstable angina
* Resting heart rate more than 120 bpm
* Resting blood pressure more than 180/100 mmHg
* Other abnormality with contribute to IMT and variable measurement

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Maximal Inspiratory pressure | "baseline, pre-intervention" and "6 weeks"
Systolic and diastolic blood pressure | "baseline, pre-intervention" and "6 weeks"
  blood pressure will include systolic and diastolic blood pressure
Six-minute walk distance | "baseline, pre-intervention" and "6 weeks"

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Phayao, Nai Muang, Changwat Phayao, Thailand

IPD SHARING:
Plan to Share IPD: No